CLINICAL TRIAL: NCT06858267
Title: The Impact of Meditation on Anxiety and Post-Operative Pain in Pediatric Patients Undergoing Urological Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Bradley Morganstern, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2254633
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Kidney Disease
Keywords: The Impact of Meditation on Anxiety and Post-Operative Pain in Pediatric Patients Undergoing Urological Surgery

STUDY DESIGN:
Intervention Model Description: Pediatric patients between the ages of 6 to 18 who will be undergoing urological surgery will be selected for this study along with their parents. Recruitment will begin in the clinic after surgery is scheduled. The patients will be also sign an informed consent form and assent. Patients and parents will be divided into two groups receiving meditation and not receiving meditation. The ideal meditation schedule will be 3-5 meditations per week for 5 minutes beginning 3 weeks before surgery. This will provide a dose-response relationship of meditation to anxiety and postoperative pain for data analysis.
  For randomization, the patients and their parents will be assigned a number, surveyed at 4-time points, and given a meditation regimen to see how anxiety is affected. The meditation regimen will be linked in a Qualtrics. The control group will only receive the questionnaire without meditation. The survey has eleven questions on a five-point scale ranging from "Not at all" to "A lot"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 study subjects with meditation (Experimental): The meditation regimen will be linked in a Qualtrics that is delivered to them via email daily. The patient and their parents will open the link, enter their assigned number, and follow the guided meditation embedded in the Qualtrics. This will track how many times and for how long the patients are following the regimen.
  The first PeSSKi (Perceived Stress Scale for Kids) questionnaire survey will be asked and sent via email after the appointment surgery is scheduled to assess anxiety. The second PeSSKi questionnaire survey will be over email at the halfway point to the surgery to see impact of meditation and anxiety levels at this point. The third questionnaire survey will be done immediately before the day of surgery in person to assess how anxious the patient is. The final questionnaire survey will be done 1 week postoperatively to assess the pain label of the patient is still in after the quantity of analgesic usage logged throughout the week.
  Interventions: Behavioral: PeSSKi questionnaire survey; Behavioral: Meditation Video
- 30 study subjects without meditation (Placebo Comparator): The control group will only receive the questionnaire without meditation.
  The first PeSSKi questionnaire survey will be asked and sent via email after the appointment where the surgery is scheduled to assess anxiety. The second PeSSKi questionnaire survey will be over email at the halfway point to the surgery to see the anxiety levels are at this point. The third questionnaire survey will be done immediately before the day of the surgery in person to assess how anxious the patient is. The final questionnaire survey will be done 1 week postoperatively to assess how much pain the patient is still in after the quantity of analgesic usage logged throughout the week. The questionnaire has eleven questions on a five-point scale ranging from "Not at all" to "A lot". The questionnaire link is given bellow:
  https://augusta.qualtrics.com/jfe/form/SV_2b2DZ9x16jY9IzQ (PeSSKi questionnaire) The control group will receive just the PeSSKi questionnaire.
  Interventions: Behavioral: PeSSKi questionnaire survey

INTERVENTIONS:
Behavioral: PeSSKi questionnaire survey — The control group will only receive the questionnaire without meditation. The PeSSKi questionnaire survey will be receive in 4 time point, First questionnaire will sent via email after the appointment for the surgery is scheduled. The second PeSSKi questionnaire survey will share via email at halfway point to the surgery. The third questionnaire survey will be done immediately before the day of surgery in person to assess how anxious the patient is. The final questionnaire survey will be done 1 week postoperatively to assess how much pain the patient is still in after the quantity of analgesic usage logged throughout the week.
Behavioral: Meditation Video — The experimental group pediatric patients selected for this study and their parents will be receiving meditation and PeSSKi (Perceived Stress Scale for Kids) questionnaire. The ideal meditation schedule will be 3-5 meditations per week for 5 minutes beginning 3 weeks before surgery. This will provide a dose-response relationship of meditation to anxiety and postoperative pain for data analysis. The Patient and their parents will open the link, enter their assigned number, and follow the guided meditation embedded in the Qualtrics. This will track how many times and for how long the patients are following the regimen.
  The questionnaire has eleven questions on a five-point scale ranging from "Not at all" to "A lot". An example of the meditation video questionnaire is linked here:
  https://augusta.qualtrics.com/jfe/form/SV_3DeFFKdJVupMJQq (experimental group) https://augusta.qualtrics.com/jfe/form/SV_2b2DZ9x16jY9IzQ (PeSSKi questionnaire)
  Arms: 30 study subjects with meditation

SUMMARY:
1. The aim of this study is to assess anxiety in pediatric patients preoperatively, perioperatively, and postoperatively and whether meditation reduces anxiety in the days before, during, and after the surgery.
2. The second aim of this study is to see if longitudinal meditation is associated with decreased postoperative pain by examining whether the group prescribed meditation has reduced pain medication intake, measured by the frequency of liquid analgesic medicine intake.

DETAILED DESCRIPTION:
Up to 70% of pediatric patients experience preoperative and perioperative anxiety. The anxiety level of their parents or guardians also affects the anxiety levels of pediatric patients themselves. Anxiety levels often peak during the time of anesthesia induction, suggesting the unfamiliar physical environment plays a role in increasing anxiety levels. Pediatric anxiety often manifests in various ways such as strong emotions, physical noncompliance, and regression. Pre-operative anxiety has been shown to increase the risk of cardiovascular events during the operation, increase difficulty gaining access to intubation, and increase anesthetic requirements. The effects of pre-operative anxiety do not end once the operation is complete. Rather, there have been suggestions that preoperative anxiety has a positive association with postoperative pain and prolonged hospital stay. Thirteen percent of pediatric surgical patients have postoperative pain that interferes with their daily activities or sleep patterns. In addition, 25-63% of pediatric patients who undergo urological surgeries experience moderate to severe pain on postoperative day 1 and the pain decreases but persists for 2 days on average. Therefore, it is worthwhile to explore noninvasive and adaptable methods to decrease preoperative anxiety among the patient and their guardians'.

Mindfulness is turning one's awareness of past and future events inward to focus on the present time. The practice provides an opportunity for people to reflect on their current internal conditions in a space and time that is not pressured, which can improve their ability to healthily and effectively respond to those conditions. One such study proposed that trait mindfulness and perceived anxiety have an inverse relationship. While another showed those with higher levels of trait mindfulness have increased resistance to stress and psychological flexibility. By embracing the entire spectrum of emotions one may encounter in the present or about a future event, people may be able to feel relief instead of increased anxiety or worry.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18
* Pediatric urology patients at Children's Healthcare of Georgia in Augusta, GA; scheduled for any urological surgery
* Otherwise, healthy patients
* Must record any medical history and medications
* Must record prior attempts of meditation therapy
* Children must provide assent

Exclusion Criteria:

* History of any prior surgeries
* History of anxiety or anxiety-related disorders
* Diagnosis of developmental delay

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Meditation may decrease preoperative anxiety among the patient and their guardians. And to see if longitudinal meditation is associated with decreased postoperative pain by examining frequency of liquid analgesic medicine intake. | Active participation in the study will last for about one month, this includes three weeks pre-operatively and one week post-operatively. Total duration of the project is approximately two years.
  Number of participants with meditation as assessed to change pain label from baseline in pain score on the scale at 1-week postoperative condition. The final questionnaire survey will be done 1 week postoperatively to assess how much pain the patient is still in after the quantity of analgesic usage logged throughout the week.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Experimental Group_ Meditation Video — https://augusta.qualtrics.com/jfe/form/SV_3DeFFKdJVupMJQq
- See also: PeSSKi (Perceived Stress Scale for Kids) questionnaire for Experimental and control group — https://augusta.qualtrics.com/jfe/form/SV_2b2DZ9x16jY9IzQ

DOCUMENTS (2):
  • Study Protocol (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT06858267/Prot_000.pdf
  • Informed Consent Form (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT06858267/ICF_001.pdf